CLINICAL TRIAL: NCT02197299
Title: Increasing Skeletal Muscle Carnitine Content to Improve Glycaemic Control in Type 2 Diabetes Mellitus
Brief Title: Improving Glycaemic Control With L-carnitine
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14/EM/0136; 13/0004659 (Other Grant/Funding Number: Diabetes UK)
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carnitine (Experimental): Oral administration of 4.5 g L-carnitine L-tartrate (containing 3 g L-carnitine; Carnipure, Lonza Ltd., Switzerland) once daily for 24 weeks
  Interventions: Dietary Supplement: L-carnitine
- Sugar pill (Placebo Comparator): Oral administration of placebo sugar pill
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-carnitine
  Arms: Carnitine
Dietary Supplement: Placebo
  Arms: Sugar pill

SUMMARY:
A characteristic of Type 2 diabetes is a high blood glucose level, which is partly caused by the inability of insulin to stimulate glucose uptake into our muscles (insulin resistance). Insulin resistance can be caused by the accumulation of fat within muscle of overweight individuals. The aim of the present research is to test whether a novel nutritional intervention containing L-carnitine can increase the amount of carnitine within muscle of individuals recently diagnosed with Type 2 diabetes. Carnitine is essential for 'burning fat' within our muscles and it is hoped that increasing the amount of carnitine within muscle can increase fat burning, lower muscle fat, reverse insulin resistance and ultimately lower blood glucose levels and wellbeing. We also aim to investigate the cellular mechanisms underlying any observed effects in a hope to identify further targets to lower muscle fat.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 27-37 kg/m2
* Male
* Age 18-60 years old
* Type 2 diabetes mellitus reasonably well controlled (HbA1c less than or equal to 58 mmol/mol) on diet therapy or metformin alone
* Not taking anti-diabetes medication other than metformin
* Understand verbal and/or written explanation of the study requirements

Exclusion Criteria:

* Malignancy (excluding localised basal and squamous cell skin cancer)
* Metabolic diseases (stable treated hypothyroidism allowed)
* Active cardiovascular disease (current angina, myocardial infarct, or coronary artery surgery/angioplasty within 12 months)
* Primary muscle disorders
* Cerebrovascular disease
* Neurological disease e.g. epilepsy, Parkinsons disease
* Active respiratory disease
* Active gastrointestinal or liver disease
* Renal impairment (eGFR <60 ml/min)
* Clotting dysfunction
* Anti-diabetes medication other than metformin
* Other medications that may affect glucose tolerance (e.g. corticosteroids), muscle metabolism, or safety (e.g. anticoagulants)
* Any other conditions in addition to the above that the investigators consider may affect study measurements or safety

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle total carnitine content | up to 24 weeks of L-carnitine supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Francis B Stephens, PhD, Principal Investigator — The University of Nottingham
Locations (1):
- David Greenfield Human Physiology Unit, School of Life Sciences, The University of Nottingham, Nottingham, United Kingdom